CLINICAL TRIAL: NCT04430582
Title: Pilot Study - Cognition in Patients With Hypoglycemia, Without Diabetes
Brief Title: Cognition in Patients With Hypoglycemia, Without Diabetes
Status: Completed | Type: Observational
Sponsor: Joslin Diabetes Center (Other)
Responsible Party: Sponsor
Other Study IDs: 00000098
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Results first posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Hypoglycemia; Cognition
Keywords: Executive Function; Memory; Post-Bariatric Hypoglycemia
MeSH Terms: conditions — Hypoglycemia | interventions — Electrocardiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hypoglycemia after gastric bypass surgery - post-bariatric hypoglycemia (PBH): Participants with PBH, recruited from the Joslin Hypoglycemia Clinic and from other hypoglycemia studies at Joslin.
  Interventions: Other: Cognitive Assessment (not diagnostic); Diagnostic Test: ECG
- Post-gastric bypass participants without a history of hypoglycemia: Participants with a history of Roux-en-Y gastric bypass, but without a diagnosis of hypoglycemia, or symptoms of hypoglycemia, recruited by advertisement flyers at postoperative surgical clinics at local hospitals (such as Brigham and Women's and Beth Israel Deaconess Hospitals), research match, and from other hypoglycemia studies at Joslin.
  Interventions: Other: Cognitive Assessment (not diagnostic); Diagnostic Test: ECG

INTERVENTIONS:
Other: Cognitive Assessment (not diagnostic) — Cognitive testing will assess premorbid intelligence, working memory and attention, verbal memory and delayed memory, executive function, and psychomotor speed.
Diagnostic Test: ECG — ECG will take place during screening visit.
  Other Names: Electrocardiogram (ECG)

SUMMARY:
The purpose of this study is to determine if there are differences in cognitive function (thinking) in individuals who have recurrent hypoglycemia (low blood sugars) following Roux-en-Y gastric bypass, compared with individuals who have also had a Roux-en-Y gastric bypass but do not have hypoglycemia.

DETAILED DESCRIPTION:
This study will test the hypothesis that a history of recurrent hypoglycemia following gastric bypass is associated with differences in cognition (thinking), by analyzing results of cognitive testing in post-gastric bypass individuals with a history of hypoglycemia as compared to those without known hypoglycemia.

This pilot study will identify cognitive domains of interest, as well as inform the development of a future battery of assessments, which could be replicated in a larger sample. Cognitive domains which will be assessed include: premorbid intelligence, memory, language, executive function, and psychomotor speed.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years of age, inclusive, at screening.
2. Willingness to provide informed consent and attend one study visit.
3. For hypoglycemia after upper GI surgery group: Males or females diagnosed with ongoing post upper GI surgery hypoglycemia, with prior episodes of neuroglycopenia, unresponsive to dietary intervention.
4. For hypoglycemia without a history of upper gastrointestinal surgery group: Males or females diagnosed with ongoing hypoglycemia with prior episodes of neuroglycopenia, and without a history of prediabetes, diabetes, or upper GI surgery.
5. For post-bariatric without hypoglycemia group: Males or females with history of bariatric surgery, and no history of symptomatic hypoglycemia.
6. For non-surgical controls only: Males or females with no history of upper GI surgery and no history of hypoglycemia, prediabetes, or diabetes.

Exclusion Criteria:

1. Active treatment with any diabetes medications, except for acarbose.
2. History of cerebrovascular accident.
3. History of a traumatic brain injury not related to hypoglycemia.
4. Active depression.
5. Active alcohol abuse or substance abuse.
6. Known insulinoma, gastrinoma or other neuroendocrine tumor.
7. Having undergone same / similar cognitive assessments within the last calendar year.

There will be no involvement of special vulnerable populations such as fetuses, neonates, pregnant women, children, prisoners, institutionalized or incarcerated individuals, or others who may be considered vulnerable populations.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited into 2 groups: (1) patients with hypoglycemia after upper gastrointestinal surgery (PBH), recruited from the Joslin Hypoglycemia Clinic, (2) asymptomatic post-bariatric patients without hypoglycemia, recruited from postoperative surgical clinics at Brigham and Women's Hospital or Beth Israel Hospitals.
  Some participants may be recruited from other hypoglycemia studies at Joslin.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2021-08-04 (Actual); Study Completion 2021-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Elizabeth Patti, MD, Principal Investigator — Joslin Diabetes Center
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Puleio A, Sheehan A, Musen G, Patti ME. Cognition in patients with post-bariatric hypoglycemia. Obesity (Silver Spring). 2024 Mar;32(3):466-471. doi: 10.1002/oby.23862. Epub 2023 Sep 5. PMID 37667837

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In August of 2020 recruitment began. Potential participants were recruited from the Joslin Diabetes Center hypoglycemia clinic, local advertisement, research match, and through participation in other studies. Recruitment ended August of 2021.
Pre-assignment Details: There were plans to include controls (no history of gastric bypass, no hypoglycemia). 3 were recruited and assessed. Upon analysis they did not match age/BMI of the post-bariatric hypoglycemia (PBH) group, and with a low number, were excluded from the design.
  3 additional participants were subsequently excluded upon review of history/records: 2 with no history of gastric bypass, and 1 with a traumatic brain injury (revealed upon detailed medical history).
Period: Overall Study
Arm/Group | Hypoglycemia After Gastric Bypass Surgery - Post-bariatric Hypoglycemia (PBH) | Post-gastric Bypass Participants Without a History of Hypoglycemia
Started | 8 | 8
Completed | 7 | 7
Not Completed | 1 | 1
Not completed — Found to meet exclusionary criteria | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hypoglycemia After Gastric Bypass Surgery - Post-bariatric Hypoglycemia (PBH) | Post-gastric Bypass Participants Without a History of Hypoglycemia | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Median (Standard Deviation); unit: years] | 56 (8) | 52 (9) | 54.5 (9.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 7 | 5 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 6 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Northeastern United States
  participants
    United States | 7 | 7 | 14
Current body mass index (kg/m^2) [Median (Standard Deviation); unit: kg/m^2] | 31.4 (5.4) | 32.9 (11.3) | 31.5 (9.575)
Body composition fat percentage (%) [Median (Standard Deviation); unit: percent] | 41.5 (11.9) | 41.5 (12.7) | 41.5 (10.5)
Patient Health Questionnaire-2 (PHQ-2) score [Median (Standard Deviation); unit: Scores on a scale (range 0 to 6)] — Patient Health Questionnaire-2 (PHQ-2) scores were used to measure depressive symptoms. Scores for this assessment range from 0 to 6, with a higher score indicating greater severity of depressive symptoms.
  Scores on a scale (range 0 to 6) | 1 (2.5) | 0 (0) | 0.5 (1.75)
Beck Depression Inventory score [Median (Standard Deviation); unit: Scores on a scale (range is 0 to 63)] — Beck Depression Inventory scores were used to measure depressive symptoms. Scores for this assessment range from 0 to 63, with a higher score indicating greater severity of depressive symptoms.
  Scores on a scale (range is 0 to 63) | 8 (9.5) | 7 (7) | 7.5 (8.2)
Alcohol Use Disorders Identification Test (AUDIT-C) score [Median (Standard Deviation); unit: Scores on a scale (range 0 to 10)] — Alcohol Use Disorders Identification Test (AUDIT-C) scores were used to measure alcohol use. Scores for this assessment range from 0 to 10, with a higher score indicating more alcohol use.
  Scores on a scale (range 0 to 10) | 0 (1.5) | 1 (1.5) | 0.5 (1.5)
Alcohol use (drinks per week) [Median (Standard Deviation); unit: number of alcoholic drinks per week] | 0 (0.25) | 0.25 (0.31) | 0.115 (0.4625)
Number of participants with a smoking history [Count of Participants; unit: Participants] | 2 | 1 | 3
Number of participants using recreational marijuana [Count of Participants; unit: Participants] | 2 | 0 | 2
Years of education [Median (Standard Deviation); unit: years] | 14 (2) | 16 (4) | 16 (2)
Duration of hypoglycemia (years) [Median (Standard Deviation); unit: years] | 3 (3.775) | 0 (0) | 3 (3.8)

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Immediate Verbal Memory
Description: Rey Auditory Verbal Learning Test (RAVLT) immediate recall accuracy scores was used to measure immediate verbal memory. Scores for this assessment were compared between groups. Scores for this assessment range 0 to 69, with a higher score indicating a superior immediate verbal memory. Wilcoxon rank-sum tests was used to examine differences between groups.
Time Frame: During the one day of cognitive assessment administration.
Measure: Median (Standard Deviation); unit: RAVLT scores on a scale (range 0 to 69)
Arm/Group | Hypoglycemia After Gastric Bypass Surgery - Post-bariatric Hypoglycemia (PBH) | Post-gastric Bypass Participants Without a History of Hypoglycemia
Number analyzed (Participants) | 7 | 7
RAVLT scores on a scale (range 0 to 69) | 50 (6) | 48 (14.5)
Statistical Analysis 1: Comparison: Hypoglycemia After Gastric Bypass Surgery - Post-bariatric Hypoglycemia (PBH) vs Post-gastric Bypass Participants Without a History of Hypoglycemia; Test type: Other; p = 0.90, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Assessment of Delayed Verbal Memory
Description: RAVLT 20 minute recall accuracy scores, was used to measure delayed memory and was compared between groups. Scores for this assessment range 0 to 15, with a higher score indicating less delays in memory. Wilcoxon rank-sum tests was used to examine differences between groups.
Time Frame: During the one day of cognitive assessment administration.
Measure: Median (Standard Deviation); unit: RAVLT scores on a scale (range 0 to 15)
Arm/Group | Hypoglycemia After Gastric Bypass Surgery - Post-bariatric Hypoglycemia (PBH) | Post-gastric Bypass Participants Without a History of Hypoglycemia
Number analyzed (Participants) | 7 | 7
RAVLT scores on a scale (range 0 to 15) | 9 (2) | 10 (1.5)
Statistical Analysis 1: Comparison: Hypoglycemia After Gastric Bypass Surgery - Post-bariatric Hypoglycemia (PBH) vs Post-gastric Bypass Participants Without a History of Hypoglycemia; Test type: Other; p = 0.24, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Working Memory Assessed by the Letter Number Sequencing Scaled Score
Description: Letter-Number Sequencing subtest from the Wechsler Memory Scale III scaled scores were used to measure working memory and were compared between groups. Wilcoxon rank-sum test was used to examine differences between groups. Scores for this assessment range 1 to 19, with a higher score indicating a superior working memory.
Time Frame: During the one day of cognitive assessment administration.
Measure: Median (Standard Deviation); unit: Scores on a scale (range 1 to 19)
Arm/Group | Hypoglycemia After Gastric Bypass Surgery - Post-bariatric Hypoglycemia (PBH) | Post-gastric Bypass Participants Without a History of Hypoglycemia
Number analyzed (Participants) | 7 | 7
Scores on a scale (range 1 to 19) | 10 (2.5) | 10 (1)
Statistical Analysis 1: Comparison: Hypoglycemia After Gastric Bypass Surgery - Post-bariatric Hypoglycemia (PBH) vs Post-gastric Bypass Participants Without a History of Hypoglycemia; Test type: Other; p = 0.74, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Assessment of Cognitive Flexibility Using Trails Scaled Score
Description: Delis-Kaplan Executive Function System (DKEFS),Trail Making Task score was used to assess the cognitive flexibility component of executive function. Scores are derived from time to complete the task plus errors. Wilcoxon rank-sum test was used to examine differences between groups. Normative scores for this assessment range 1-19 (mean of 10, and standard deviation of 3), and a higher score indicates superior cognitive flexibility.
Time Frame: During the one day of cognitive assessment administration.
Measure: Median (Standard Deviation); unit: Scores on a scale (range 1 to 19)
Arm/Group | Hypoglycemia After Gastric Bypass Surgery - Post-bariatric Hypoglycemia (PBH) | Post-gastric Bypass Participants Without a History of Hypoglycemia
Number analyzed (Participants) | 7 | 7
Scores on a scale (range 1 to 19) | 12 (2) | 11 (1.5)
Statistical Analysis 1: Comparison: Hypoglycemia After Gastric Bypass Surgery - Post-bariatric Hypoglycemia (PBH) vs Post-gastric Bypass Participants Without a History of Hypoglycemia; Test type: Other; p = 0.51, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Assessment of Cognitive Flexibility Using Color-word Inference Test
Description: DKEFS Color-Word Interference Test (CWIT) Inhibition Switching scores was used to measure the cognitive flexibility component of executive function. The CWIT is scored by time to complete plus errors. Wilcoxon rank-sum test was used to examine differences between groups. Normative scores for this assessment range 1-19 (mean of 10, and standard deviation of 3), and a higher score indicates superior cognitive flexibility.
Time Frame: During the one day of cognitive assessment administration.
Measure: Median (Standard Deviation); unit: Scores on a scale (range 1 to 19)
Arm/Group | Hypoglycemia After Gastric Bypass Surgery - Post-bariatric Hypoglycemia (PBH) | Post-gastric Bypass Participants Without a History of Hypoglycemia
Number analyzed (Participants) | 7 | 7
Scores on a scale (range 1 to 19) | 11 (1.5) | 12 (3.5)
Statistical Analysis 1: Comparison: Hypoglycemia After Gastric Bypass Surgery - Post-bariatric Hypoglycemia (PBH) vs Post-gastric Bypass Participants Without a History of Hypoglycemia; Test type: Other; p = 0.70, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Assessment of Inhibition Using Color-word Inference Test
Description: DKEFS CWIT scores was used to measure the inhibition component of executive function. The CWIT is scored by time to complete plus errors. Wilcoxon rank-sum test was used to examine differences between groups. Normative scores for this assessment range 1-19 (mean of 10, and standard deviation of 3), and a higher score indicates superior inhibition.
Time Frame: During the one day of cognitive assessment administration.
Measure: Median (Standard Deviation); unit: Scores on a scale (range 1 to 19)
Arm/Group | Hypoglycemia After Gastric Bypass Surgery - Post-bariatric Hypoglycemia (PBH) | Post-gastric Bypass Participants Without a History of Hypoglycemia
Number analyzed (Participants) | 7 | 7
Scores on a scale (range 1 to 19) | 10 (2) | 11 (4)
Statistical Analysis 1: Comparison: Hypoglycemia After Gastric Bypass Surgery - Post-bariatric Hypoglycemia (PBH) vs Post-gastric Bypass Participants Without a History of Hypoglycemia; Test type: Other; p = 0.95, Kruskal-Wallis

7. Secondary Outcome: Verbal Ability Cognitive Control Assessed by Letter Fluency
Description: DKEFS Letter Fluency Task will be used to assess the verbal functioning cognitive control ability component of executive function. Scores are derived from the number of unique, correct words. Wilcoxon rank-sum test was used to examine differences between groups. Normative scores for this assessment range 1-19 (mean of 10, and standard deviation of 3), and a higher score indicates superior verbal functioning cognitive control ability.
Time Frame: During the one day of cognitive assessment administration.
Measure: Median (Standard Deviation); unit: Scores on a scale (range 1 to 19)
Arm/Group | Hypoglycemia After Gastric Bypass Surgery - Post-bariatric Hypoglycemia (PBH) | Post-gastric Bypass Participants Without a History of Hypoglycemia
Number analyzed (Participants) | 7 | 7
Scores on a scale (range 1 to 19) | 8 (3.5) | 12 (2)
Statistical Analysis 1: Comparison: Hypoglycemia After Gastric Bypass Surgery - Post-bariatric Hypoglycemia (PBH) vs Post-gastric Bypass Participants Without a History of Hypoglycemia; Test type: Other; p = 0.48, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Assessment of Psychomotor Speed
Description: The grooved pegboard test is a manipulative dexterity task that assesses psychomotor speed, fine motor control, and rapid-visual motor coordination. Participants were asked to insert 25 grooved pegs into holes within the given time limit up to 300 seconds (the score upper limit is thus 300). Time taken to complete the test has been found to be inversely correlated with cognitive ability; therefore, a higher score represents an inferior score. Wilcoxon rank-sum test was used to examine differences between groups.
Time Frame: During the one day of cognitive assessment administration.
Measure: Median (Standard Deviation); unit: Seconds
Arm/Group | Hypoglycemia After Gastric Bypass Surgery - Post-bariatric Hypoglycemia (PBH) | Post-gastric Bypass Participants Without a History of Hypoglycemia
Number analyzed (Participants) | 7 | 7
Seconds | 100 (10.5) | 102 (15)
Statistical Analysis 1: Comparison: Hypoglycemia After Gastric Bypass Surgery - Post-bariatric Hypoglycemia (PBH) vs Post-gastric Bypass Participants Without a History of Hypoglycemia; Test type: Other; p = 0.85, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Verbal Ability Cognitive Control Assessed by Category Fluency
Description: DKEFS Category Fluency scores were used to measure cognitive control of verbal ability, specifically measuring an individuals ability to access and retrieve semantic information (memory) as a component of executive function. Category fluency is scored by number of correct words plus errors in a 60 second trial in each of 3 categories. Wilcoxon rank-sum test was used to examine differences between groups. Normative scores for this assessment range 1-19 (mean of 10, and standard deviation of 3), and a higher score indicates superior cognitive control of verbal ability.
Time Frame: During the one day of cognitive assessment administration.
Measure: Median (Standard Deviation); unit: Scores on a scale (range 1 to 19)
Arm/Group | Hypoglycemia After Gastric Bypass Surgery - Post-bariatric Hypoglycemia (PBH) | Post-gastric Bypass Participants Without a History of Hypoglycemia
Number analyzed (Participants) | 7 | 7
Scores on a scale (range 1 to 19) | 10 (3) | 14 (1)
Statistical Analysis 1: Comparison: Hypoglycemia After Gastric Bypass Surgery - Post-bariatric Hypoglycemia (PBH) vs Post-gastric Bypass Participants Without a History of Hypoglycemia; Test type: Other; p = 0.01, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Verbal Ability Cognitive Flexibility, Assessed by Category Switching Scaled Score
Description: DKEFS Category Switching scores will be used to measure cognitive control of verbal ability, specifically measuring an individuals ability to access and retrieve semantic information (memory), switching back and forth between 2 different semantic categories, a component of executive function. Category switching is scored by number of correct words plus errors. Wilcoxon rank-sum test was used to examine differences between groups. Normative scores for this assessment range 1-19 (mean of 10, and standard deviation of 3), and a higher score indicates superior cognitive control of verbal ability.
Time Frame: During the one day of cognitive assessment administration.
Measure: Median (Standard Deviation); unit: Scores on a scale (range 1 to 19)
Arm/Group | Hypoglycemia After Gastric Bypass Surgery - Post-bariatric Hypoglycemia (PBH) | Post-gastric Bypass Participants Without a History of Hypoglycemia
Number analyzed (Participants) | 7 | 7
Scores on a scale (range 1 to 19) | 10 (2) | 15 (4.5)
Statistical Analysis 1: Comparison: Hypoglycemia After Gastric Bypass Surgery - Post-bariatric Hypoglycemia (PBH) vs Post-gastric Bypass Participants Without a History of Hypoglycemia; Test type: Other; p = 0.01, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Verbal Ability Cognitive Control of Inhibition, Assessed by Category Switching Accuracy Scaled Score
Description: DKEFS Category Switching Accuracy scores will be used to measure cognitive control of verbal ability, specifically measuring an individuals ability to inhibit incorrect or repetitive semantic information (memory), while switching back and forth between 2 different semantic categories, a component of executive function. Wilcoxon rank-sum test was used to examine differences between groups. Normative scores for this assessment range 1-19 (mean of 10, and standard deviation of 3), and a higher score indicates superior cognitive control of verbal ability.
Time Frame: During the one day of cognitive assessment administration.
Measure: Median (Standard Deviation); unit: Scores on a scale (range 1 to 19)
Arm/Group | Hypoglycemia After Gastric Bypass Surgery - Post-bariatric Hypoglycemia (PBH) | Post-gastric Bypass Participants Without a History of Hypoglycemia
Number analyzed (Participants) | 7 | 7
Scores on a scale (range 1 to 19) | 10 (2) | 14 (3)
Statistical Analysis 1: Comparison: Hypoglycemia After Gastric Bypass Surgery - Post-bariatric Hypoglycemia (PBH) vs Post-gastric Bypass Participants Without a History of Hypoglycemia; Test type: Other; p = 0.03, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Lexical Processing Assessed by Letter Fluency, First Interval.
Description: DKEFS Letter Fluency, first interval scores will be used to measure cognitive control of lexical processing, specifically measuring an individuals ability to retrieve phonemic information, a component of executive function. Participants are asked to name as many words a they are able starting with a specific letter, without repetition. Wilcoxon rank-sum test was used to examine differences between groups. There are four intervals of this task the first assessing initiation of retrieval while the following trials measuring the ability to sustain retrieval. Normative scores for this assessment range 1-19 (mean of 10, and standard deviation of 3), and a higher score indicates superior cognitive control of lexical processing.
Time Frame: During one day of cognitive assessement administration.
Measure: Median (Standard Deviation); unit: Scores on a scale (range 1 to 19)
Arm/Group | Hypoglycemia After Gastric Bypass Surgery - Post-bariatric Hypoglycemia (PBH) | Post-gastric Bypass Participants Without a History of Hypoglycemia
Number analyzed (Participants) | 7 | 7
Scores on a scale (range 1 to 19) | 10 (3.5) | 13 (3)
Statistical Analysis 1: Comparison: Hypoglycemia After Gastric Bypass Surgery - Post-bariatric Hypoglycemia (PBH) vs Post-gastric Bypass Participants Without a History of Hypoglycemia; Test type: Other; p = 0.03, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Lexical Processing as Assessed by Letter Fluency, Second Interval
Description: DKEFS Letter Fluency, second interval scores will be used to measure cognitive control of lexical processing, specifically measuring an individuals ability to retrieve phonemic information, a component of executive function. There are four intervals of this task the second through fourth trial assess ability to sustain retrieval. Participants are asked to name as many words a they are able starting with a specific letter, without repetition. Wilcoxon rank-sum test was used to examine differences between groups. Normative scores for this assessment range 1-19 (mean of 10, and standard deviation of 3), and a higher score indicates superior cognitive control of lexical processing.
Time Frame: During one day of cognitive assessement administration.
Measure: Median (Standard Deviation); unit: Scores on a scale (range 1 to 19)
Arm/Group | Hypoglycemia After Gastric Bypass Surgery - Post-bariatric Hypoglycemia (PBH) | Post-gastric Bypass Participants Without a History of Hypoglycemia
Number analyzed (Participants) | 7 | 7
Scores on a scale (range 1 to 19) | 10 (5) | 11 (2)
Statistical Analysis 1: Comparison: Hypoglycemia After Gastric Bypass Surgery - Post-bariatric Hypoglycemia (PBH) vs Post-gastric Bypass Participants Without a History of Hypoglycemia; Test type: Other; p = 0.30, Wilcoxon (Mann-Whitney)

14. Secondary Outcome: Lexical Processing Assessed by Letter Fluency, Third Interval
Description: DKEFS Letter Fluency, third interval scores will be used to measure sustainment of cognitive control of lexical processing, specifically measuring an individuals ability to continue to retrieve phonemic information after multiple trials, a component of executive function. There are four intervals of this task the second through fourth trial assess ability to maintain retrieval. Participants are asked to name as many words a they are able starting with a specific letter, without repetition. Wilcoxon rank-sum test was used to examine differences between groups. Normative scores for this assessment range 1-19 (mean of 10, and standard deviation of 3), and a higher score indicates superior sustainment of cognitive control of lexical processing.
Time Frame: During one day of cognitive assessment administration.
Measure: Median (Standard Deviation); unit: Scores on a scale (range 1 to 19)
Arm/Group | Hypoglycemia After Gastric Bypass Surgery - Post-bariatric Hypoglycemia (PBH) | Post-gastric Bypass Participants Without a History of Hypoglycemia
Number analyzed (Participants) | 7 | 7
Scores on a scale (range 1 to 19) | 10 (1.5) | 12 (2)
Statistical Analysis 1: Comparison: Hypoglycemia After Gastric Bypass Surgery - Post-bariatric Hypoglycemia (PBH) vs Post-gastric Bypass Participants Without a History of Hypoglycemia; Test type: Other; p = 0.045, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: Lexical Processing Assessed by Letter Fluency, Fourth Interval
Description: DKEFS Letter Fluency, fourth interval scores will be used to measure sustainment of cognitive control of lexical processing, specifically measuring an individuals ability to continue to retrieve phonemic information after multiple trials, a component of executive function. There are four intervals of this task the second through fourth trial assess ability to maintain retrieval. Participants are asked to name as many words a they are able starting with a specific letter, without repetition. Wilcoxon rank-sum test was used to examine differences between groups. Normative scores for this assessment range 1-19 (mean of 10, and standard deviation of 3), and a higher score indicates superior sustainment of cognitive control of lexical processing.
Time Frame: During one day of cognitive assessment administration.
Measure: Median (Standard Deviation); unit: Scores on a scale (range 1 to 19)
Arm/Group | Hypoglycemia After Gastric Bypass Surgery - Post-bariatric Hypoglycemia (PBH) | Post-gastric Bypass Participants Without a History of Hypoglycemia
Number analyzed (Participants) | 7 | 7
Scores on a scale (range 1 to 19) | 8 (6) | 11 (1.5)
Statistical Analysis 1: Comparison: Hypoglycemia After Gastric Bypass Surgery - Post-bariatric Hypoglycemia (PBH) vs Post-gastric Bypass Participants Without a History of Hypoglycemia; Test type: Other; p = 0.37, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the single study visit for each participant.
Arm/Group | Hypoglycemia After Gastric Bypass Surgery - Post-bariatric Hypoglycemia (PBH) | Post-gastric Bypass Participants Without a History of Hypoglycemia
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

LIMITATIONS AND CAVEATS:
Limitations of this pilot study include its small sample size, cross-sectional approach, and low power (increased risk of type 2 error).

The battery of tests utilized was specifically limited to maintain a total assessment time of no more than one hour, in order to reduce the impact of participant fatigue.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-18): https://cdn.clinicaltrials.gov/large-docs/82/NCT04430582/Prot_SAP_000.pdf